CLINICAL TRIAL: NCT00862901
Title: A Phase I Trial of Continuous Low-Irradiance Photodynamic Therapy (CLIPT) for Patients Failing Radiation Therapy
Brief Title: Safety Study Using Photodynamic Therapy Light Therapy for Patients With Chest Wall Progression of Breast Cancer and Satellite Metastases of Melanoma
Acronym: CLIPT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); Axcan Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Komen Award ID# -BCTR0707871; Komen Award ID# -BCTR0707871; IRB # 8227
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Breast Cancer; Skin Cancer
Keywords: cancer; skin metastases; chest wall progression of breast cancer; malignant melanoma; photodynamic therapy; photophrin; satellite and in-transit metastases of malignant melanoma; skin cancer
MeSH Terms: conditions — Breast Neoplasms; Skin Neoplasms; Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): 100 J / cm2 over 24 hours
  Interventions: Device: CLIPT patch
- 2 (Experimental): 200 J / cm2 over 24 hours
  Interventions: Device: CLIPT patch
- 3 (Experimental): 400 J / cm2 over 24 hours
  Interventions: Device: CLIPT patch
- 4 (Experimental): 800 J / cm2 over 24 hours
  Interventions: Device: CLIPT patch

INTERVENTIONS:
Device: CLIPT patch — A Diomed laser will deliver 630nm (red spectrum) light through a Fiber optic Patch. The Fiber Optic Patch will be compatible with the laser, delivering light to a designated region on the patient's skin. Patients will receive a single intravenous injection of Photofrin (0.8mg/kg body weight) 36 - 48 hours prior to the CLIPT procedure. PDT will be delivered over 24 hours for the dose of each arm. Patients will be enrolled in sequential cohorts of six, at increasing laser intensity until the maximum tolerated dose is reached.

SUMMARY:
This research is intended to explore a new approach to therapy when breast cancer recurs in the skin. The treatment, known as continuous low-irradiance photodynamic therapy, or CLIPT, has shown great promise in animal studies. The investigators goal is to evaluate CLIPT in people, using a novel light delivery system, to assess its side effects and the benefit it has in treating cancer. The investigators goal is to develop a safe, effective therapy that can be given in the doctor's office or possibly at home.

DETAILED DESCRIPTION:
The goal of this research is to conduct a Phase I clinical study to assess the toxicity, safety and feasibility of a novel cancer treatment, Continuous Low Irradiance Photodynamic Therapy (CLIPT). This research will provide translation of recent promising preclinical work to human subjects with recurrent breast cancer.

BACKGROUND: Patients who develop post-mastectomy chest wall skin recurrence and fail conventional radiation therapy have few therapeutic options that can result in durable control. High-irradiance photodynamic therapy (PDT) has shown efficacy in patients with chest-wall progression of breast cancer that have failed radiation, surgery, and chemotherapy. However its clinical application has been severely limited as currently employed methods of PDT result in virtually 100% of patients develop skin necrosis, large areas of full-thickness ulceration, slow healing and chronic wound pain. In the rat and rabbit-brain tumor models, reducing the laser irradiance and increasing the exposure time to achieve a similar total fluence (fluence = irradiance x time) to standard PDT, avoids tissue necrosis while inducing apoptosis in the tumor but not normal tissue.

HYPOTHESIS: Low dose-rate (low irradiance) PDT may reduce or eliminate skin toxicity and enables treatment of skin/subcutaneous chest wall metastases in skin previously subjected to ionizing radiation.

SPECIFIC AIMS:

1) determine the fluence of CLIPT resulting in toxicity (maximum tolerated dose), defined as ulceration or necrosis of previously irradiated skin (non-tumor bearing skin within the prior ionizing radiation field) or normal skin, 2) evaluate the feasibility, ergonomics and safety of performing CLIPT via a proprietary electronically targetable fiber-optic "patch" placed directly on tumor-bearing, surrounding uninvolved previously irradiated skin and normal integument 3) study the tumor-bearing integument for clinical response to therapy by measuring complete, partial and no response to CLIPT.

STUDY DESIGN: We will perform a standard dose (laser fluence) escalation trial (holding drug level constant) in human subjects with post-mastectomy skin recurrences that have failed ionizing radiation therapy and assess toxicity in previously irradiated and normal integument.

POTENTIAL OUTCOMES & BENEFITS: Therapeutic options for post-mastectomy cutaneous recurrences failing conventional radiotherapy are limited. If the pre-clinical results are replicated in human subjects, Phase II studies to evaluate CLIPT would be warranted. The long-term goal is to develop an unobtrusive, large-area CLIPT system in the form of a fiber-optically woven "garment" that can be worn by the patient outside the hospital setting for repeated and extended periods without causing skin breakdown or pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age, with primary or metastatic cutaneous tumors that have been previously irradiated.
* Patients must have a target lesion and normal peri-umbilical skin that can be covered by the fiber-optic mesh used to deliver CLIPT (10 x 10 cm for Target lesion, and 1 x 1 cm for Control site).
* Patients must have a target lesion in a location other than the hands, feet, genitals, or face. Lesions in those locations will be excluded.
* Patients must sign informed consent.

Exclusion Criteria:

* Patients must not have received any systemic anti-cancer therapy within 30 days prior to enrolling in this study.
* Patients must not have received radiation therapy to the target site within 60 days of enrolling on this study.
* Patients with medical conditions associated with photosensitivity, such as cutaneous porphyria or a collagen vascular disease, or with known allergies to porphyrins will be excluded.
* Pregnant and nursing patients will be excluded. Women of child-bearing potential must have a negative serum or urine pregnancy test prior to enrollment.
* Patients taking medications known to cause photosensitivity (tetracyclines, sulfonamides, phenothiazines, sulfonylurea hypoglycemic agents, thiazide diuretics, griseofulvin, and fluoroquinolones) will be excluded.
* Laboratory values (Note: these are provided by the potential patient):
* Absolute neutrophil count > 1000.
* Patients with severe hepatic dysfunction (total bilirubin, AST, or ALT > five times upper limit of normal) will be excluded.
* Adequate coagulation status as indicated by platelet count > 50,000, PT and PTT < 1.5 time the upper limit of normal.
* Negative Urine or Serum Pregnancy Test

Note: No cost to patient, and no compensation provided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (full thickness ulceration and/or necrosis of the skin) | 48 hours to 7 days after treatment

SECONDARY OUTCOMES:
Efficacy and mechanism of action of CLIPT. | 24 hours after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roger Graham, MD, Principal Investigator — Tufts Medical Center, Department of Surgery
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States